CLINICAL TRIAL: NCT00965120
Title: The Effect of Ischaemic-Reperfusion in Man - A Bradykinin Dependent Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Aarhus (Other); University of Oxford (Other)
Responsible Party: Christian M Pedersen, clinical research fellow, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CMP 3
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Ischaemic Heart Diseases
Keywords: Ischaemia reperfusion; Bradykinin; Platelet activation; Endothelial function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Bradykinin Receptor Antagonists; icatibant; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Ischaemia 20 minutes. Blood pressure cuff will be inflated to 200mmHg around the upper arm for 20 minutes to induce ischaemia. Systemic infusion of placebo (saline).
  Interventions: Procedure: Forearm vascular study; Drug: Placebo (saline)
- 2 (Active Comparator): Ischaemia 20 minutes. Blood pressure cuff will be inflated to 200mmHg around the upper arm for 20 minutes to induce ischaemia. Systemic infusion of bradykinin receptor antagonist (HOE-140).
  Interventions: Procedure: Forearm vascular study; Drug: bradykinin receptor antagonist (HOE-140)

INTERVENTIONS:
Procedure: Forearm vascular study — Forearm blood flow measured by venous occlusion plethysmography during interarterial infusion of vasodilators (Ach). Venous blood sampling via cannula in antecubital fossa.
Drug: bradykinin receptor antagonist (HOE-140) — Systemic infusion of bradykinin receptor antagonist (HOE-140).
  Arms: 2
Drug: Placebo (saline) — Systemic infusion of placebo (saline).
  Arms: 1

SUMMARY:
Heart attacks are usually caused by a blood clot blocking an artery supplying blood to the heart. Current treatments are designed to relieve this blockage as quickly as possible to minimize damage to the heart muscle. However in restoring the supply of blood local damage known as "ischaemia-reperfusion injury" may occur. The aim of this study is to assess how clot forming and clot dissolving pathways are affected during this process, and examine the role of a natural inflammatory hormone, bradykinin. This will help the investigators to understand the mechanism by which ischaemia-reperfusion injury may occur and to devise new treatments for heart attacks.

ELIGIBILITY:
Inclusion Criteria:

* healthy males between 18-65 years of ages
* non-smokers

Exclusion Criteria:

* any concurrent illness or chronic medical condition
* concurrent use of vasoactive medication
* smoking history

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow in response to vasodilators (ACh) and ischaemia reperfusion | 20 fixed timepoints during each study visit (3hrs)

SECONDARY OUTCOMES:
Change in platelet-monocyte-binding after ischaemia reperfusion | 4 fixed timepoints during each study visit (3hrs)

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Study Director — University of Edinburgh; Rajesh K Kharbanda, PhD, FRCP, Study Director — University of Oxford
Locations (1):
- University of Edinburgh, 49 Little France Crescent, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Pedersen CM, Schmidt MR, Barnes G, Botker HE, Kharbanda RK, Newby DE, Cruden NL. Bradykinin does not mediate remote ischaemic preconditioning or ischaemia-reperfusion injury in vivo in man. Heart. 2011 Nov;97(22):1857-61. doi: 10.1136/heartjnl-2011-300323. Epub 2011 Aug 26. PMID 21873443